CLINICAL TRIAL: NCT04764578
Title: Sexual Dysfunction Following Upper Extremity Trauma
Status: Withdrawn | Type: Observational
Why Stopped: Staffing shortages
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jed Maslow, Assistant Professor, Department of Orthopaedic Surgery, Vanderbilt University Medical Center
Other Study IDs: 210352
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Sexual Dysfunction; Upper Extremity Trauma
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis

1. The prevalence of sexual dysfunction after upper extremity function in adults (>18yo) is higher than the general population in the early post-operative period (3mo) and at 1 year post-operatively.
2. Null: Adult patients (<18 yo) with isolated upper extremity trauma do not experience sexual dysfunction more than the general population.

Primary Study Question

a) What is the prevalence of sexual dysfunction after upper extremity trauma (fracture, soft tissue disruption, neurovascular injury, and completion amputation) in adult patients?

Secondary Study Questions

1. Are there patient or injury factors that can predict sexual dysfunction?
2. Do certain fractures cause more sexual dysfunction than others?
3. Can we accurately predict which patients may experience sexual dysfunction post-injury?

DETAILED DESCRIPTION:
Enrollment Visit Following the consent process, patient demographics, injury information, and baseline pre-trauma sexual function will be documented as part of the patient's baseline assessment. Participants will be asked to complete the study survey which will combine 1 question (Item 21 Sexual Dysfunction) from the Disabilities of Arm, Shoulder and Hand (DASH) and the 5 question, Likert-like, Arizona Sexual Experience Scale (ASEX)7,8 . Depending on the participant's response to survey item 1, they may or may not be asked to complete the remaining 5 questions. As part of routine care in the Department of Orthopaedics, patients being seen in the Hand & Upper Extremity outpatient clinics are asked to complete the following surveys: QuickDASH, SANE, PROMIS Physical Function CAT and PROMIS Anxiety CAT. The study will access/utilize the responses to these routine care patient reported outcomes to correlate to our study survey responses. This routine care PRO data will be stored in the electronic health record. Project team members listed as Key Study Personnel with existing electronic health record (EHR) system access rights may be granted use of REDCap Clinical Data Interoperability Services (CDIS) tools. These tools are designed to enable transfer of relevant study-related data from the Vanderbilt Research Derivative and/or directly from the EHR into REDCap. If KSP are unable to transfer data using CDIS, it will be manually entered into the REDCap database. If, for some reason, the participant does not complete the routine care PROs at their enrollment visit, we will ask them to complete the surveys as part of the study.

Follow-up Visits Participants will be asked to complete the same study survey at their 3 month, 6 month and 12 month follow-up visits. The study will access/utilize the routine care PRO responses (QuickDASH, SANE, PROMIS Physical Function CAT and PROMIS Anxiety CAT) at these visits, also. If, for some reason, the participant does not complete the routine care PROs at their follow-up visit, we will ask them to complete the surveys as part of the study.

If the participant does not have a routine care appointment scheduled at the follow-up visit time points, misses a routine care follow-up appointment or the study staff are not available to collect data at these follow-up appointments, the research coordinator will attempt to contact the patient by phone, mail or electronically using REDCap, to obtain the outcomes data.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > 18 years old with an isolated upper extremity injury treated operatively or non-operatively at Vanderbilt University Medical Center
* Isolated upper extremity is defined as:
* Fractures, stratified by level
* Hand (phalanx, metacarpal), wrist (carpal, distal radius), forearm (radial shaft, ulnar shaft, both bone), elbow (distal humerus, proximal ulna, radial head), arm (humeral shaft), shoulder (proximal humerus, scapula, clavicle)
* Soft tissue trauma involving ligament or muscle injury requiring repair or soft tissue defect requiring flap coverage
* Nerve injury, stratified by level
* Peripheral nerve injury vs plexus injury
* Vascular injury
* Amputation
* Combined injury

Exclusion Criteria:

* Age < 18 at time of injury
* Traumatic brain injury
* Other concomitant orthopaedic injury to the lower extremities
* Other trauma requiring hospital admission (abdominopelvic, thoracic, head or spine trauma)
* Patients with bilateral upper extremity injuries

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be identified when they present to Vanderbilt University Medical Center or Vanderbilt Department of Orthopaedic Clinics for follow up for their isolated upper extremity trauma.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (Item 21 Sexual Dysfunction) Score | Change between baseline, 3-month, 6-month, and 12-month visits.
  The DASH item response ranges from 1 (no difficulty) to 5 (unable).
  21 Item Sexual Dysfunction from the Disabilities of Arm, Shoulder and Hand (DASH)
Arizona Sexual Experience Scale (ASEX) Score | Change between baseline, 3-month, 6-month, and 12-month visits.
  The Arizona Sexual Experience Scale (ASEX) is a 5 item Likert-like scale with response ranges from 1 (extremely easily) to 6 (never).